CLINICAL TRIAL: NCT06854211
Title: Mechanisms of Opioid-induced Respiratory Depression (OIRD) During Sleep
Brief Title: Impacts of Opioids on Respiratory Drive During Sleep
Acronym: OIRD
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Danny J. Eckert, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2024P002115
Record Dates: First submitted 2025-02-18; First posted 2025-03-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Opioids; Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Morphine (Active Comparator)
  Interventions: Drug: Morphine p.o.
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine p.o. — Morphine 50mg PO will be given on sleep study night.
  Arms: Morphine
Drug: Placebo — Placebo will be given on the sleep study night.
  Arms: Placebo

SUMMARY:
The investigators are studying the impact that opioids have on breathing during sleep in healthy participants and those diagnosed with obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy controls: Apnea Hypopnea Index (AHI) < 5 events/hr on in-laboratory PSG within 3 months of enrollment
* OSA group: AHI > 10 events/hr on in-laboratory PSG within 3 months of enrollment; treated or untreated.

Exclusion Criteria:

* Sleep disordered breathing or respiratory disorders (other than OSA in the OSA group), such as central sleep apnea (>50% of respiratory events scored as central), chronic hypoventilation/hypoxemia (awake SaO2 < 92% by oximetry) due to chronic obstructive pulmonary disease or other respiratory conditions.
* Other sleep disorders: periodic limb movements (periodic limb movement index > 20/hr), narcolepsy, or parasomnias.
* Any unstable major medical condition.
* Medications expected to stimulate or depress respiration (including other opioids taken at home, barbiturates, benzodiazepines, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* History of allergy to lidocaine or oxymetazoline.
* Contraindications for morphine, including:
* allergy to morphine or opioids
* chronic obstructive pulmonary disease, asthma, or other significant respiratory disorders
* kidney or liver dysfunction, as this can affect the metabolism and excretion of morphine, leading to increased risk of toxicity.
* women who are pregnant or breastfeeding will be excluded due to potential risks to the fetus or infant.
* history of substance abuse, particularly opioid abuse, will be excluded to prevent potential misuse or relapse.
* current use of central nervous system depressants.
* individuals with gastrointestinal obstruction. Constipation is not an exclusion criterion because morphine is only administered for one night.
* recent head injury, brain tumors, or other conditions leading to increased intracranial pressure.
* unstable heart disease, particularly those with risk factors for or a history of heart rhythm disorders.
* epilepsy or a history of seizures, as morphine can lower the seizure threshold.
* severe psychiatric conditions, particularly those with a history of psychosis, as opioids can exacerbate these conditions.
* medications that interact with morphine, such as selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants (TCAs), Monoamine oxidase inhibitors (MAOIs), and the atypical antidepressants buproprion and trazodone.
* untreated or unstable endocrine disorders like adrenal insufficiency or thyroid dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The change in ventilation (L) per minute during stable sleep with morphine versus placebo. | From enrollment to the end of treatment at 6 weeks.
  The primary outcome, determining the change in ventilation in liters per minute, will be analyzed on both subpopulations (controls and people with obstructive sleep apnea) using generalized linear mixed models with treatment, period and sequence as fixed effects and a random effect of participant nested within sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Danny J Eckert, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.